CLINICAL TRIAL: NCT04870684
Title: Interest of Thromboelastometry as a Biomarker of Post-thrombolysis or Post-thrombectemia Revascularization Success in Ischemic Stroke: a Prospective, Single-center, Observational Study in an Emergency Department
Brief Title: Thromboelastometry and Ischemic Stroke (ThromboPredict)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A00171-40
Record Dates: First submitted 2021-04-09; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Cerebrovascular Stroke; Thrombolytic Therapy; Mechanical Thrombectomy
Keywords: thromboelastometry; ischemic stroke; biomarker; thrombolysis; endovascular thrombectomy; Prediction of revascularization
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sucess of revascularization: group of patients for whom after thrombolysis neurological improvement will be observed and recanalization on imaging will be seen.
  Interventions: Other: thromboelastometry test

INTERVENTIONS:
Other: thromboelastometry test — This study does not modify the usual care of the patient. Only 5 citrated tubes (maximum 15 mL of blood) are collected in addition to the initial emergency department sample (routine care). The patient's care follows the classic thrombolysis alert pathway. There is no additional complementary examination or additional neurological evaluation. Clot formation kinetics will be evaluated by thromboelastometry to determine the predictive parameters of revascularization. Clot formation and lysis parameters as well as revascularization according to thrombo-inflammation processes will be studied.

SUMMARY:
In ischemic stroke, the recanalization rate after intravenous thrombolysis has been estimated to be less than 50% in patients with proximal intracranial artery occlusion; this rate is greater than 80% after endovascular thrombectomy. Thromboelastometry is a method of analysis of coagulation and fibrinolysis in whole blood. The main objective of this study is to evaluate whether the parameters obtained by thromboelastometry are predictive of revascularization at arteriography during mechanical thrombectomy, after treatment with rt-PA thrombolysis.

DETAILED DESCRIPTION:
This is a single-center prospective observational study at the University Hospital of Caen. Any patient presenting a neurological deficit of sudden onset, compatible with a ischemic stroke diagnosed on brain imaging and eligible for thrombolysis by rtPA and/or a endovascular thrombectomy procedure will be included. Clot formation kinetics will be assessed by thromboelastometry (ROTEM® and/or QUANTRA®) to determine the predictive parameters of revascularization. The parameters of clot formation and lysis as well as revascularization according to thrombo-inflammation processes will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of ischemic stroke
* Decision of intravenous thrombolysis and/or endovascular thrombectomy by the neurologist and/or interventional neuroradiologist.
* Patient admitted to the emergency department during the hours and days when the hematology-biology laboratory is open (Monday to Friday from 8:30 a.m. to 6:30 p.m.)
* No opposition to the research from the patient or his relatives
* Inclusions according to the emergency procedure

Exclusion Criteria:

* Age < 18 ans
* Formal contraindication to thrombolysis and/or endovascular thrombectomy, disorders of hemostasis and anticoagulant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years with a diagnosis of ischemic stroke compatible and eligible for intravenous thrombolysis (IVT) with rt-PA and/or endovascular thrombectomy (EVT).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of the success of the revascularization procedure by thromboelastometry | One hour after the blood test
  All the parameters of clot formation and lysis will be studied, in particular the area under the curve (AUC)
Does clot firmness could predict the success of the revascularization | One hour after the blood test
  clot firmness (MCF in millimeter, mm)
Prediction of the success of the revascularization procedure by thromboelastometry | One hour after the blood test
  clot lysis time (seconde).

SECONDARY OUTCOMES:
Thomboelastometry and prediction of thrombolysis + thrombectomy efficacy | during thrombectomy procedure
  effectiveness of thrombectomy will be assessed per-arteriogram by the TICI score (Grade 0: no perfusion Grade 1: penetration with minimal perfusion Grade 2: partial perfusion Grade 2A: only partial filling (less than two-thirds) of the entire vascular territory is visualized Grade 2B: complete filling of all of the expected vascular territory is visualized but the filling is slower than normal Grade 3: complete perfusion)
Thomboelastometry and prediction of thrombectomy efficacy | immediatly after thrombectomy procedure
  number of passes required for successful recanalization thrombolysis
Thomboelastometry and prediction of thrombectomy efficacy | through study completion, an average of 3 years
  puncture to recanalization (minute)
Thomboelastometry and prediction of success of recanalization by thrombectomy alone | just at the end of thrombectomy procedure
  Effectiveness of thrombectomy will be assessed by the TICI score ((Grade 0: no perfusion Grade 1: penetration with minimal perfusion Grade 2: partial perfusion Grade 2A: only partial filling (less than two-thirds) of the entire vascular territory is visualized Grade 2B: complete filling of all of the expected vascular territory is visualized but the filling is slower than normal Grade 3: complete perfusion)
Prediction of success of thrombolysis | "Day 1", "Day 3" after thrombolysis
  presence or absence of a clot on MRI or angioscan
Thomboelastometry and prediction of neurological outcome | "D0", "Day 1", "Day 3" after revascularization
  The use of the NIHSS score will allow the neurological evaluation of the patient (at admission and 24h/72h after the recanalization attempt). Neurological outcome, as assessed by the NIHSS score, is considered favorable if the NIHSS score at 24h/72h post-recanalization is equal to 0 or 1 or if there is an improvement in the NIHSS score of at least four points between the admission score and the score at 24h/72h post-recanalization.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Macrez, Doctor, Principal Investigator — University hospital of Caen and faculty of medicine
Locations (1):
- University hospital of Caen, emergency department, Caen, France

IPD SHARING:
Plan to Share IPD: Yes
Sample and clinical could be share with private researcher (STAGO)
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: At the end of the inclusion period
Access Criteria: The clinical and biological databases will be recorded by investigators and laboratory biologists respectively from the existing hospital information system. Anonymized data will be transferred via a secure server and encrypted messaging